CLINICAL TRIAL: NCT03105154
Title: Experience With the Negative Pressure Incision Management System (Prevena) in Vascular Surgery Patients With High Risk for Groin Wound Infection
Brief Title: Groin Wound Infection Rate Using Prevena Compared to Standard Dressing in Vascular Surgery Patients With High Risk
Acronym: PREVENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Levester Kirksey, MD, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-1402
Record Dates: First submitted 2017-03-14; First posted 2017-04-07 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Endovascular Procedures

STUDY DESIGN:
Intervention Model Description: Patient will be randomized sequentially to Prevena alternating with standard of care dressing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevena Dressing (Experimental): Groin dressed with Prevena
  Interventions: Other: Prevena Dressing
- Conventional Dressing (Active Comparator): Groin dressed with conventional bandage
  Interventions: Other: Conventional Dressing

INTERVENTIONS:
Other: Prevena Dressing — Prevena dressing is applied on one groin
  Arms: Prevena Dressing
Other: Conventional Dressing — Conventional dressing is applied on the contralateral groin
  Arms: Conventional Dressing

SUMMARY:
Evaluate wound healing using Prevena compared to standard dressings in high risk patients after vascular surgery.

DETAILED DESCRIPTION:
Patients submitted to bilateral femoral endarterectomy will have one groin dressed with PrevenaTM and the contralateral one dressed with conventional bandage immediately after suture. Both PrevenaTM and the conventional bandage at the contralateral side will be removed before the patient discharge. Groin wound complications such as deep space infection, cutaneous cellulitis, dehiscence or re-interventions for wound-related complications will be observed in a 30-day evaluation window. This observation will be performed during the patient admission and in the post-operative standard of care visits among the first 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known bilateral vascular peripheral disease who are being evaluated for possible bilateral femoral endarterectomy
* Patients with one or more risk factor (diabetes mellitus, Obesity, heavy smoker, immunodeficiency disease, groin reoperation, prosthetic)
* Patients in follow-up at Clinic in the Vascular Surgery Department
* Sign of informed consent
* English speaking

Exclusion Criteria:

* Refusal to participate
* pregnancy
* unilateral femoral endarterectomy
* subjects for whom Prevena IMS is contraindicated

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
% of infection at 30 days | 30 days
  % of wound occurrence in the Prevena treated groin compared to conventional treated groin

CONTACTS AND LOCATIONS:
Overall Officials: Leveser Kirksey, Principal Investigator — The Cleveland Clinic
Locations (1):
- Clevealnd Clnic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No